CLINICAL TRIAL: NCT06844409
Title: Assessment of Long-Term Chemotherapy-Induced Peripheral Neuropathy and Its Impact on Quality of Life in Colon Cancer Patients After Neoadjuvant Platinum-Containing Chemotherapy
Brief Title: Neoadjuvant FOLFOX Chemotherapy for Colon Cancer: Long-Term Chemotherapy-Induced Peripheral Neuropathy and Impact on Quality of Life
Acronym: NEOCIPN-COLON
Status: Completed | Type: Observational
Sponsor: P. Herzen Moscow Oncology Research Institute (Other Government)
Collaborators: Jiaxing University (Unknown)
Responsible Party: Principal Investigator, Yulia Karagodina, Researcher, P. Herzen Moscow Oncology Research Institute
Other Study IDs: 72-2021
Record Dates: First submitted 2025-02-07; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN)
Keywords: chemotherapy-induced peripheral neuropathy; oxaliplatin; quality of life; neoadjuvant chemotherapy; colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with colon cancer (II-III stage) who received neoadjuvant FOLFOX chemotherapy: 54 Patients with locally advanced colon cancer who received platinum-containing chemotherapy as the initial phase of their treatment, followed by surgical resection and, if indicated, adjuvant chemotherapy

SUMMARY:
The goal of this observational study was to learn about the long-term effects of neoadjuvant (pre-surgery) chemotherapy on patients with locally advanced colon cancer. The main focus was to better understand the severity of long-lasting nerve damage, known as chemotherapy-induced peripheral neuropathy (CIPN), and its impact on patients' quality of life (QoL).

The key question the study aimed to answer was: What is the long-term severity of this common adverse event, and how much of an impact does it have on patients' quality of life?

Participants provided detailed responses about the severity of their CIPN symptoms and the overall impact on their well-being using the FACT-GOG-Ntx questionnaire.

DETAILED DESCRIPTION:
Introduction. Chemotherapy-induced peripheral neuropathy (CIPN) is a common and debilitating side effect experienced by many cancer patients receiving neurotoxic agents such as oxaliplatin. CIPN can manifest as numbness, tingling, and neuropathic pain, significantly impairing patients' quality of life (QoL). While the acute development of CIPN during chemotherapy treatment is well documented, the long-term persistence and severity of CIPN symptoms after completion of therapy is less understood.

The relatively new approach to treatment of patients with locally advanced colon cancer involves starting treatment with neoadjuvant (pre-operative) chemotherapy regimens containing oxaliplatin, such as FOLFOX, followed by definitive surgical resection and potentially additional adjuvant chemotherapy. This strategy has proven to be non-inferior to more established adjuvant (post-operative) chemotherapy, according to results of several clinical trials. However, the impact of this long-term CIPN on patient-reported outcomes and QoL in the setting of neoadjuvant chemotherapy has not been thoroughly investigated.

Additionally, there is interest in exploring whether modifying the sequence of neoadjuvant and adjuvant chemotherapy regimens could potentially mitigate the severity of CIPN. Specifically, a hypothesis can be made that delivering a reduced volume of oxaliplatin-containing chemotherapy (6 cycles of neoadjuvant FOLFOX) followed by a break for surgery, with only selective use of additional adjuvant chemotherapy based on response, may result in less cumulative neurotoxicity and improved long-term CIPN outcomes compared to the standard approach of administering the full course of chemotherapy after surgery.

The primary objective of this observational study was to characterize the long-term severity of CIPN symptoms and the associated impact on QoL in patients with locally advanced colon cancer who received neoadjuvant FOLFOX chemotherapy, followed by surgical resection and response-dependent adjuvant chemotherapy.

Study Design and Participants. This was a single-center, prospective observational study conducted at an academic medical center. Adult patients (≥18 years old) with histologically confirmed, locally advanced adenocarcinoma of the colon (clinical stage III or high-risk stage II) were eligible for enrollment. Key inclusion criteria included an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, adequate organ function, and no prior systemic chemotherapy or radiotherapy.

Eligible patients were enrolled and received 6 cycles of neoadjuvant FOLFOX chemotherapy. FOLFOX consisted of oxaliplatin 85 mg/m2 IV on day 1, leucovorin 400 mg/m2 IV on day 1, and 5-fluorouracil 400 mg/m2 IV bolus on day 1 followed by 2400 mg/m2 continuous IV infusion over 46 hours, every 2 weeks.

After completing six cycles of neoadjuvant FOLFOX chemotherapy, patients underwent definitive surgical resection of their primary tumor. For those who achieved a favorable pathologic response (defined as pT0-2N0M0 or pT3N0M0 without risk factors), no additional adjuvant chemotherapy was administered post-surgery. However, in cases of pT3N0M0 with the presence of risk factors, patients received 3 months of adjuvant capecitabine. Patients with a poor pathologic response were offered an additional six cycles of adjuvant FOLFOX chemotherapy.

Assessment of CIPN. Throughout the course of treatment, patients underwent clinical assessments for the development of CIPN. During treatment, a physician performed a neurological examination and graded the severity of CIPN using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0. This standardized grading system classifies CIPN from grade 1 (mild) to grade 4 (life-threatening).

At a minimum of 3 months after the end of platinum-containing chemotherapy treatment, patients completed the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT-GOG-Ntx) questionnaire. The FACT-GOG-Ntx is a validated, patient-reported outcome measure that evaluates the severity of CIPN symptoms and their impact on daily functioning and QoL.

The primary endpoint of this observational study was assessment of the long-term severity of CIPN and its impact on QoL, as measured by the FACT-GOG-Ntx questionnaire. The secondary target was assessment of correlation between various risk factors (older age (> 65 years), diabetes, Eastern Cooperative Oncology Group (ECOG) performance status, Body mass index (BMI) > 25, and higher cumulative oxaliplatin dose; cold temperatures during treatment) and severity of long-term CIPN.

Statistical Considerations. Descriptive statistics were used to summarize characteristics of patients. Associations between risk factors and ACIPN severity were evaluated using chi-squared tests. Two-tailed Mann-Whitney U tests were used to show significant differences in long-term CIPN outcomes and QoL scores between patient groups. Pearson and Spearman correlations were used to evaluate associations between risk factors and CIPN severity. Statistical significance was set at p < 0.05. Statistical analyses were performed using JASP (Version 0.18.3), an open-source statistical software package (JASP Team, 2024) or GraphPad Prism (GraphPad Software, San Diego, CA, USA).

Results. Between March 2021 and February 2024, a total of 54 patients were included and assessed by clinicians for acute CIPN during treatment. 45 of these patients provided complete FACT-GOG-Ntx questionnaire data for the long-term CIPN assessment, and 40 were included in the QoL analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, histologically confirmed, resectable colon cancer stage IIA - IIIC (cT3N0M0 [depth of invasion > 5 mm], cT4a-T4bN0M0, T1-4N1-2M0).
* Age < 75 years.
* ECOG performance status 0-1.
* Hemoglobin > 9 g/dL.
* Absolute neutrophil count > 1500/µL.
* Platelet count > 100,000/µL.
* Bilirubin level < 1.5 times the upper limit of normal.
* Creatinine clearance > 60 mL/min (calculated using the Cockcroft-Gault formula).
* ALT and AST levels < 2.5 times the upper limit of normal.

Exclusion Criteria:

* Presence of distant metastases.
* History of other oncological diseases, except for:

  1. Cured non-melanoma skin cancer without known signs of recurrence or progression for > 5 years.
  2. Cured carcinoma in situ without signs of recurrence or progression for > 5 years.
* Clinically significant concomitant cardiac pathology (chronic heart failure NYHA class > 1; hypertension with a risk of cardiovascular complications > 3; history of myocardial infarction, stroke, or transient ischemic attack; presence of other decompensated cardiovascular diseases).
* ECOG performance status > 1.
* Presence of viral or infectious diseases (human immunodeficiency virus, chronic viral hepatitis, other infectious diseases in the acute phase).
* History of clinically significant central nervous system disorders.
* Clinically significant peripheral polyneuropathy (> grade 2).
* Pregnancy or lactation.
* Individual intolerance to the components of the treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients who were treated for locally advanced colon cancer in P. Hertsen Oncology Clinical Research Institute in Moscow, Russian Federation
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Severity of long-term chemotherapy-induced peripheral neuropathy | At least 3 months after the end of platinum-containing treatment
  Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity-13 Version 4 (FACT/GOG-Ntx) questionnaire. The FACT/GOG-Ntx total score ranges from 0-160 with higher scores indicating better QoL and/or fewer symptoms.
Patients' quality of life | At least 3 months after the end of platinum-containing treatment
  Assessment using the the Functional Assessment of Cancer Therapy-General (FACT-G) scores within the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity-13 Version 4 (FACT/GOG-Ntx) questionnaire. The FACT-G score ranges from 0-108 with higher scores indicating better QoL and/or fewer symptoms.

SECONDARY OUTCOMES:
Severity of acute chemotherapy-induced peripheral neuropathy | Through platinum-containing chemotherapy treatment completion, an average of 3,5 months
  Assessed by physicians using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0. Grading criteria for peripheral sensory neuropathy was used (grade 1-4). Higher grade indicates worse symptoms.
Correlation between risk factors and severity of chemotherapy-induced peripheral neuropathy | Through study completion, an average of 2 years
  Correlation between previously descriped risk factors (older age [> 65 years], diabetes, Eastern Cooperative Oncology Group [ECOG] performance status, Body mass index [BMI] > 25 and higher cumulative oxaliplatin dose) and severity of acute and long-term chemotherapy-induced peripheral neuropathy severity
Correlation between severity of long-term chemotherapy induced neuropathy and quality of life | At least 3 months after the end of platinum-containing treatment
  Correlation between severity of long-term chemotherapy-induced peripheral neuropathy and patients' quality of life, as assessed by Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity-13 Version 4 (FACT/GOG-Ntx) questionnaire. FACT/GOG-Ntx total score ranges from 0-160 with higher scores indicating better QoL and/or fewer symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- P. Hertsen Moscow Oncology Research Institute, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement

REFERENCES:
- [Background] Teng C; Venkatesha; Blinman PL, Vardy JL. Patterns of Patient-Reported Chemotherapy-Induced Peripheral Neuropathy in Colorectal Cancer Survivors. J Natl Compr Canc Netw. 2022 Dec;20(12):1308-1315. doi: 10.6004/jnccn.2022.7050. PMID 36509075
- [Background] Land SR, Kopec JA, Cecchini RS, Ganz PA, Wieand HS, Colangelo LH, Murphy K, Kuebler JP, Seay TE, Needles BM, Bearden JD 3rd, Colman LK, Lanier KS, Pajon ER Jr, Cella D, Smith RE, O'Connell MJ, Costantino JP, Wolmark N. Neurotoxicity from oxaliplatin combined with weekly bolus fluorouracil and leucovorin as surgical adjuvant chemotherapy for stage II and III colon cancer: NSABP C-07. J Clin Oncol. 2007 Jun 1;25(16):2205-11. doi: 10.1200/JCO.2006.08.6652. Epub 2007 Apr 30. PMID 17470850
- [Background] Soveri LM, Lamminmaki A, Hanninen UA, Karhunen M, Bono P, Osterlund P. Long-term neuropathy and quality of life in colorectal cancer patients treated with oxaliplatin containing adjuvant chemotherapy. Acta Oncol. 2019 Apr;58(4):398-406. doi: 10.1080/0284186X.2018.1556804. Epub 2019 Jan 14. PMID 30638100
- [Background] Morton D, Seymour M, Magill L, Handley K, Glasbey J, Glimelius B, Palmer A, Seligmann J, Laurberg S, Murakami K, West N, Quirke P, Gray R; FOxTROT Collaborative Group. Preoperative Chemotherapy for Operable Colon Cancer: Mature Results of an International Randomized Controlled Trial. J Clin Oncol. 2023 Mar 10;41(8):1541-1552. doi: 10.1200/JCO.22.00046. Epub 2023 Jan 19. PMID 36657089
- [Background] Davey MG, Amir AH, Ryan OK, Donnelly M, Donlon NE, Regan M, Meshkat B, Nugent E, Joyce M, Hogan AM. Evaluating the oncological safety of neoadjuvant chemotherapy in locally advanced colon carcinoma: a systematic review and meta-analysis of randomised clinical trials and propensity-matched studies. Int J Colorectal Dis. 2023 Jul 11;38(1):193. doi: 10.1007/s00384-023-04482-x. PMID 37432559